CLINICAL TRIAL: NCT05351996
Title: Does Kinesiotaping Effective for Knee Osteoarthritis? Randomized Controlled Trial
Brief Title: Kinesiotaping in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeniz Akçay, University of Health Sciences Bozyaka Training and Research Hospital Physical Medicine and Rehabilitation Department, Assoc. Prof., Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/09/2019-06
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee osteoarthritis; Kinesiotape; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Active Comparator): The participants received kinesiotape to the rectus femoris muscle.
  Interventions: Device: Kinesiotape; Other: Home-based exercise program
- Sham-kinesiotape (Sham Comparator): Non-specific taping was applied.
  Interventions: Device: Sham-kinesiotape; Other: Home-based exercise program

INTERVENTIONS:
Device: Kinesiotape — The participants received kinesiotape application three times with one-week intervals. Y strip tape was used. The interventionist applied the band to the rectus femoris muscle with facilitation technique.
  Arms: Kinesiotape
Device: Sham-kinesiotape — The participants received sham-kinesiotape application three times with one-week intervals.
  In the sham group, the interventionist adhered KT to the rectus femoris transversely, without stretching.
  Arms: Sham-kinesiotape
Other: Home-based exercise program — Participants were taught exercise program training. The exercise intervention was based on quadriceps and knee flexor muscle group strengthening, and knee joint range of motion exercises, in their home.

SUMMARY:
Kinesiotape is one of the treatment choices for the patients with knee osteoarthritis. Unlike the brace, it seems to be an important advantage in kinesiotape application in that it permits the movement of the joint. However, kinesiotape is conditionally recommended for knee osteoarthritis in the 2019 American College of Rheumatology treatment recommendations due to limiting the quality of evidence, using various application methods, and the lack of blindness concerning its use is not possible.

The aim of the study is to determine the effects of kinesiotaping on pain, physical performance, knee range of motion, and postural stability in knee osteoarthritis.

DETAILED DESCRIPTION:
Non-pharmacological treatments are recommended as first-line management in knee osteoarthritis. Kinesiotape was regarded as a supplementary intervention for patients with knee osteoarthritis. Although the results are conflicting, regarding knee osteoarthritis, recently published studies indicate beneficial effects of kinesiotape on knee-related health status, pain, quadriceps muscle strength, and range of motion. On the other hand, the measurements were performed immediately following taping or within a short-term period. The inconsistency of the study data still indicates that the efficacy of kinesiotape in knee osteoarthritis should be evaluated in randomized controlled trials. Therefore a study that investigates both short and long-term follow-up results are warranted.

This study aimed to determine the immediate and long-term effects of the single and repetitive application of kinesiotape on pain, knee joint range of motion, postural stability, and physical performance in participants with knee osteoarthritis. The results of this study will support evidence-based reports based on the effectiveness of kinesiotape in knee osteoarthritis and recommendations for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Pain for a minimum of 3 months
* Pain intensity within the last week minimum of 3 according to the visual analogue scale (VAS) at the symptomatic knee
* Grade 2-3 knee OA according to the Kellgren and Lawrence Scale
* Ability to perform the tests

Exclusion Criteria:

* Fragile, very sensitive skin, or lesions in the area
* Inflammatory arthritis
* Inability to perform functional tests
* Pregnancy
* Use of drugs associated with a psychiatric disorder
* Previous joint replacement surgery for knee/hip joints
* Diagnosis with balance disorder
* Disorders that may cause loss of muscle strength in the lower extremities
* Previous experience with the Kinesiotaping method

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As the pain intensity and pain threshold may be effected by the gender differences, the enrolled participants were consisted of females.
Enrollment: 57 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain intensity-rest at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week, 7th week
  Pain intensity was assessed by using the Visual Analogue Scale (VAS). Each patient was asked to indicate pain intensity during rest at each assessment point (on a 0-10 points numerical pain rating scale; higher scores indicate severe pain).
Change from Baseline Pain intensity-activity at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  Pain intensity was assessed by using the Visual Analogue Scale (VAS). Each patient was asked to indicate pain intensity during 50-meter walking test at each assessment point (on a 0-10 points numerical pain rating scale; higher scores indicate severe pain).

SECONDARY OUTCOMES:
Change from Baseline Knee-Related Health Status at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  To determine the baseline and the degree of change in knee-related health status Western Ontario and McMaster Universities Osteoarthritis Index was applied. Western Ontario and McMaster Universities Osteoarthritis Index, is a widely valid and reliable outcome measurement scale in patients with knee osteoarthritis. The scale consists of 24 items and is divided into three dimensions; pain; stiffness, and functionality.
Change from Baseline Pain-free Knee Range of Motion at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  Active pain-free knee range of motion examination was performed by a 360̊ double-armed universal goniometer. Knee active flexion range of motion angle without pain was measured in the supine position while the axis of the goniometer was on the femur's lateral epicondyle. For active knee extension range of motion, the investigator recorded the angle that which the participant extends the knee as much as possible. If there was an inability to reach the 0-degree starting position, the angle was given a negative value reflecting the angle missing from the full extension. Three assessment was performed and the mean value was recorded as active flexion and extension angle.
Change from Baseline Physical Function at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  The physical function of the participants enrolled in the study was evaluated by the 50-meter walking test will the subjects walk 2.5 return journeys between two cones placed 10 m apart along a walking course. The participants stood beside the cone. They were instructed to walk to the other when signaled by the investigator, go around it to the outer side, and walk back again as fast as possible.
  The time taken the task completed assessed by the same chronometer was recorded
Change from Baseline Static Postural Stability at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  The quantitative measure of the balance and postural stability of participants was performed by the Biodex Balance System (BBS). Participants completed three trial repetitions before static balance tests. For the static balance test, the participants were asked to stand with two legs on the center of the locked platform of the BBS. Three evaluations were performed in each measurement session and a mean score was calculated from the three trials. The device provides three postural stability indices (PSI) obtained by calculating the standard deviations of the degrees of an inclination concerning the zero point: overall static postural stability index (sPSI_O), static anteroposterior postural stability index (sPSI_AP), and static mediolateral postural stability index (sPSI_ML).
Change from Baseline Dynamic Postural Stability at 1st hour, 3rd week, and 7th week | Baseline (week 0), 1st hour, 3rd week , 7th week
  The quantitative measure of the balance and postural stability of participants was performed by the Biodex Balance System (BBS). Participants completed three trial repetitions before dynamic balance tests.
  During the dynamic balance test, the platform moves simultaneously to the anteroposterior (AP), or mediolateral (ML) directions in 12 different stability levels (level 1 is the least stable; level 12 is the most stable level within a 20-degree range of inclination). Dynamic PSI (dPSI) represents the variance of foot platform displacement in degrees, from level, in all motions during the test. A high number is indicative of a lot of movement during the test. Dynamic balance test was performed on the most stable level with the following parameters: duration: 20 seconds, stability level: 12, and stance: two legs

CONTACTS AND LOCATIONS:
Overall Officials: Nesibe Doğan, MD, Principal Investigator — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Hayriye Yılmaz, MSc, PT, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Buğra İnce, MD, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Şeniz Akçay, Assoc. Prof., Study Director — University of Health Sciences Izmir Bozyaka Training and Research Hospital
Locations (1):
- University of Health Sciences Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] Donec V, Kubilius R. The effectiveness of Kinesio Taping(R) for mobility and functioning improvement in knee osteoarthritis: a randomized, double-blind, controlled trial. Clin Rehabil. 2020 Jul;34(7):877-889. doi: 10.1177/0269215520916859. Epub 2020 May 6. PMID 32372651
- [Background] Kaya Mutlu E, Mustafaoglu R, Birinci T, Razak Ozdincler A. Does Kinesio Taping of the Knee Improve Pain and Functionality in Patients with Knee Osteoarthritis?: A Randomized Controlled Clinical Trial. Am J Phys Med Rehabil. 2017 Jan;96(1):25-33. doi: 10.1097/PHM.0000000000000520. PMID 27149590
- [Background] Wageck B, Nunes GS, Bohlen NB, Santos GM, de Noronha M. Kinesio Taping does not improve the symptoms or function of older people with knee osteoarthritis: a randomised trial. J Physiother. 2016 Jul;62(3):153-8. doi: 10.1016/j.jphys.2016.05.012. Epub 2016 Jun 16. PMID 27320828
- [Background] Cho HY, Kim EH, Kim J, Yoon YW. Kinesio taping improves pain, range of motion, and proprioception in older patients with knee osteoarthritis: a randomized controlled trial. Am J Phys Med Rehabil. 2015 Mar;94(3):192-200. doi: 10.1097/PHM.0000000000000148. PMID 25706053